CLINICAL TRIAL: NCT01562951
Title: cAlprotectin and hsCRP as Markers of a New Diagnostic-therapeutic strAtegy That Assesses muCosal Activity to individuaLize Treatment and Improve the Prognosis of Patients With Crohn's Disease Treated With Immunosuppressants
Brief Title: Assessment of Mucosal Activity to Improve the Prognosis of Patients With Crohn's Disease Treated With Immunosuppressants
Acronym: ADACAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not enough patient population according to selection criteria to complete the study
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Collaborators: Abbott (Industry); TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A12-771
Record Dates: First submitted 2012-03-13; First posted 2012-03-26 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Crohn's Disease; Mucosal Inflammation
Keywords: Crohn's disease; mucosal inflammation; lesions
MeSH Terms: conditions — Crohn Disease; Mucositis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLACEBO (Placebo Comparator): Treatment with placebo
  Interventions: Drug: Placebo
- ADALIMUMAB (Active Comparator): Treatment with Adalimumab
  Interventions: Drug: ADALIMUMAB

INTERVENTIONS:
Drug: ADALIMUMAB — Adalimumab at 160/80 mg and maintained on 40 mg eow until next colonoscopy performed at week 48. If before week 48, an increase of more than 50% is observed in calprotectin and/or hsCRP from baseline, over two consecutive follow up visits 2 weeks apart, the colonoscopy will be performed earlier. If patients have still significant endoscopic lesions, adalimumab or adalimumab placebo will be intensified to 40 mg weekly.
  Other Names: HUMIRA
  Arms: ADALIMUMAB
Drug: Placebo — PLACEBO at 160/80 mg and maintained on 40 mg eow until next colonoscopy performed at week 48. If before week 48, an increase of more than 50% is observed in calprotectin and/or hsCRP from baseline, over two consecutive follow up visits 2 weeks apart, the colonoscopy will be performed earlier. If patients have still significant endoscopic lesions, adalimumab or adalimumab placebo will be intensified to 40 mg weekly
  Arms: PLACEBO

SUMMARY:
This study will test that individualized treatment in patients with Crohn's Disease in remission or mild clinical activity under immunosuppressants may improve prognosis, rather than just treating flares.

DETAILED DESCRIPTION:
Patients will be prescreened for inclusion criteria one week before the start of screening at Visit 0 (Prescreening Visit). Patients must be on stable doses of azathioprine/mercaptopurine. Patients will be given a diary to record their CD symptoms for the seven days prior to Visit 1. At Visit 1 (Screening Visit 1), patients will have their CDAI score assessed based upon their diary information. Patients with CDAI ≤ 220 will then have both calprotectin and hsCRP testing done. Patients with calprotectin > or = 250µg/g and/or hsCRP > or = 5mg/L will be notified and told to schedule Visit 2 within three weeks. At Visit 2 (Screening Visit 2), patients will undergo a colonoscopy. A Crohn's Disease Endoscopic Index of Severity (CDEIS) will be used to determine the endoscopic activity. Patients with significant endoscopic lesions will be notified and asked to enroll in the study.

Patients will be randomized into the study at Visit 3 (Randomization Visit, same day of Visit 2 in results available). Due to the cost and invasiveness of the colonoscopy, the Screening Visit 2 colonoscopy will serve as the baseline for the study, should the patient be enrolled. Drug will also be dispensed at this visit. Eligible patients will be randomized in a 1:1 ratio to receive either adalimumab or placebo during the treatment period, along with continuing their current immunosuppressive maintenance treatment at a stable dose. Treatment in both arms will be induction at 160/80mg and maintenance on 40 mg every other week.

Patients will return for follow up visits every 12 weeks until the final follow-up visit at 48 weeks (Visit 7), where another colonoscopy will be performed. Patients who terminate early from the study for any reason will be asked to return for a follow-up visit, where Visit 7 procedures will be performed.

Before week 48, if a patient has an increase of more than 50% in either calprotectin and/or hsCRP over baseline and above the thresholds at any regular visit, a follow-up visit will be performed two weeks later. If the 50% increase is still observed another colonoscopy will be performed, within two weeks of the follow-up visit. If patients still have significant endoscopic lesions, study product will be intensified to 40 mg weekly. This will include patients on placebo in order to preserve the double-blind aspect of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old- Patients with CD diagnosis confirmed by colonoscopy
* Patients with inflammatory CD of terminal ileal, colonic or ileocolonic location
* Maintenance treatment with at least 2 mg/kg/day for azathioprine/ 1 mg/kg/day for mercaptopurine or the highest dosage tolerated in patients who could not tolerate this dosage, at least 6 months.
* Willingness to sign informed consent
* If female of childbearing age, be post-menopausal, surgically sterile, or willing to use a reliable form of birth control for the duration of the study (such as physical barrier [patient and partner], contraceptive pill or patch, spermicide and barrier, or intrauterine device)and for at least five months after the last adalimumab treatment.
* Able to comply with the requirements of the study.
* CDAI score ≤ 220.
* Calprotectin > or = 250µg/g and/or hsCRP > or = 5mg/L.
* Significant lesions seen during colonoscopy, as defined by CDEIS.

Exclusion Criteria:

* Patients with an ostomy, or ileoanal pouch (subject with previous ileo-rectal anastomosis are not excluded), draining fistula, abscess
* Patients who had intestinal resection within one year.
* Symptomatic stricture either diagnosed by colonoscopy or clinically suspected and confirmed by imaging techniques.
* Prior treatment with any anti-tumor necrosis factor (TNF) drug.
* Patients receiving rectal treatment 1 month before inclusion
* Signs of active infection
* Previous history of active untreated or inadequately treated tuberculosis (TB) or latent TB. Patients should be screened for latent TB as per local guidelines or clinical practice in the country of study conduct. Patients with latent TB should be treated with standard antimycobacterial therapy (for at least 4 weeks) before initiating biologic therapy and have a negative CRX for active TB at screening
* Subjects with a poorly controlled medical condition such as: uncontrolled diabetes with documented history of recurrent infections, unstable ischemic heart disease, moderate to severe congestive heart failure (New York Heart Association [NYHA] class III or IV), recent cerebrovascular accident, or any other condition which, in the opinion of the Investigator or the sponsor, would put the subject at risk by participation in the protocol
* Signs of colon cancer or dysplasia
* Signs of severe or unstable renal, hepatic, gastrointestinal, cardiovascular, respiratory, neurological, psychiatric, or hematological disease
* Signs of cancer in the past five years, except for localized and treated basal cell skin cancer or cervical cancer
* Patients who are pregnant or nursing
* Concomitant treatment with:

  * Live vaccines.
  * 5-ASA compounds: Rectal 5-ASA should be discontinued at least 4 weeks before study inclusion. Oral 5-ASA must be at a stable dose for at least 4 weeks before study inclusion. If oral 5-ASA has recently been discontinued, 4 weeks should pass before study inclusion.
  * Oral corticosteroids (eg., Prednisone, budesonide) should be discontinued for 3 months before study inclusion.
  * Antibiotics for CD. Only antibiotics used to treat a concurrent infection are allowed.
  * Immunomodulators:

Patients receiving therapy with azathioprine/mercaptopurine must have been on a stable dose for at least 12 weeks before inclusion and must continue with the same dose during the study.

No treatment with other known immunomodulators (eg. methotrexate, 6-thioguanine [6-TG], cyclosporine, tacrolimus, sirolimus, ustekinumab, pentoxifylline, or mycophenolate mofetil) or experimental drugs (eg., factor colony stimulating granulocyte macrophage [GM-CSF]) within 6 months

* Monoclonal antibodies or anti-TNF drugs.
* Aspirin or Non-steroidal anti-inflammatory drugs (NSAIDs). Treatment with aspirin and/or NSAIDS should not occur for more than 15 consecutive days before collecting of the stool sample for Calprotectin and performing the colonoscopy.

  - Screening laboratory and other analyses show any of the following abnormal results:
* Aspartate transaminase (AST) or alanine transaminase (ALT) > 2 x the upper limit of the reference range;
* Total bilirubin ≥ 3 mg/dL (51 μmol/L);
* Serum creatinine > 1.6 mg/dL (144 μmol/L)

  * History of any drug or alcohol abuse in the past 2 years
  * Receipt of other study product within 3 months of inclusion in this study
  * Patients employed by the sponsor or in any relationship of dependence with the sponsor and/or investigator
  * Staff at the study center
  * Hypersensitivity to the active substance or to any of the excipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the rate of therapeutic failure up to week 48 | Every 12 weeks up to Week 48
  The therapeutic failure is defined as any of following cases:
  1. CDAI > 220 with at least 70-point increase from baseline over two consecutive visits 12 weeks apart or CDAI > 300 at any time point during the study;
  2. need of any change in therapy for CD except the ones planned per protocol in each group of the study;
  3. need of surgery related to CD or of stricture endoscopic dilatation.

SECONDARY OUTCOMES:
The rate of therapeutic failure (see the definition of primary endpoint) up to week 24 | up to week 24
Change in CDEIS from baseline to week 48 | up to week 48
  CDEIS = Crohn's Disease Endoscopic Index of Severity.
The rate of mucosal healing (CDEIS=0) at week 48 | at week 48
  CDEIS = Crohn's Disease Endoscopic Index of Severity
The rate of CDEIS remission (CDEIS<=3) at week 48 | at week 48
  CDEIS = Crohn's Disease Endoscopic Index of Severity
The rate of CDEIS response, which is defined as a decrease of at least 4 points in CDEIS from baseline to week 48 | from baseline up to week 48
  CDEIS = Crohn's Disease Endoscopic Index of Severity
Change in CDAI from baseline to week 12, 24, 36 and 48 | from baseline to week 12, 24, 36 and 48
  CDAI = Crohn's Disease Activity Index.
Change in the global score based on IBDQ from baseline to week 12, 24, 36, and 48. | from baseline to week 12, 24, 36, and 48.
  IBDQ = Inflammatory Bowel Disease Questionnaire.
Area Under the Curve (AUC) over 48 weeks for CDAI | 48 weeks
The number of surgical interventions related to CD up to 24 and 48 weeks | up to 24 and 48 weeks
The rate of hospital admissions related to the disease, to the treatment side effects or other causes up to weeks 24 or 48 | up to weeks 24 or 48
The rate of serious AEs between the two strategies up to 24 and 48 weeks | up to 24 and 48 weeks
The rate of serious AEs requiring the cessation of the ongoing treatment between the two strategies up to 24 and 48 weeks. | up to 24 and 48 weeks
The accuracy of calprotectin/hsCRP to predict therapeutic failure 12 weeks in advance | 12 weeks
The correlation between calprotectin, hsCRP and CDAI at any time points during the study. | 48 weeks
  Pearson Product-Moment Correlation will be used to evaluate correlations between calprotectin, hsCRP and CDAI at all scheduled visits.
The correlation between calprotectin/hsCRP and CDEIS or mucosal healing at Baseline and Week 48. | at Baseline and Week 48.
  Pearson Product-Moment Correlation will also be used to evaluate between calprotectin (and hsCRP) and CDEIS at Baseline and Week 48.
Change in the scores based on WPAI from baseline to week 12, 24, 36 and 48 | from baseline to week 12, 24, 36 and 48
  WPAI = Work Productivity and Activity Impairment Questionnaire
The change in calprotectin and hsCRP from baseline to week 12, 24, 36, and 48 | from baseline to week 12, 24, 36, and 48

CONTACTS AND LOCATIONS:
Overall Officials: VALLE GARCÍA, MD, Principal Investigator — Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa
Locations (30):
- Belgium (6):
  - Imeldaziekenhuis Bonheiden, Bonheiden, Bonheiden
  - Hospital Erasme Bruxelles, Brussels, Brussels Capital
  - Hospital Saint Luc Bruxelles, Brussels, Brussels Capital
  - Hospital University Gent, Ghent, Gent
  - Centre Hospitalier Universitaire de Liege, Liège, Liege
  - Heiling Hartzieknhuis Roeselare, Roeselare, Roeselare
- France (12):
  - CHU Amiens - Hospital Nord, Amiens, Amiens
  - CHU Bordeaux - Hospital Haut-Leveque, Pessac, Bordeaux
  - Hospital Beaujon, Clichy, Clichy
  - CHRU Lille - Hospital Claude Huriez, Lille, Lille
  - CHU Lyon Sud, Lyon, Lyon
  - CHU Nancy - Hospital de Brabois Adultes, Vandœuvre-lès-Nancy, Nancy
  - CHU Nantes, Nantes, Nantes
  - Hospital Saint Louis, Paris, Paris
  - CHRU Reims - Hospital Robert Debre, Reims, Reims
  - CHU Rouen - Hospital Charles Nicolle, Rouen, Rouen
  - CH Saint Etienne - Hospital Nord, Saint-Etienne, Saint Etienne
  - CHU Tours - Hospital Trousseau, Chambray, Tours
- Spain (12):
  - Complejo Hospitalario Santiago de Compostela, Santiago de Compostela, A coruña
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Doctor Negrin, Las Palmas de Gran Canarias, Canary Islands
  - Hospital Universitario La Princesa, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Virgen del Rocío, Seville, Sevilla
  - Hospital de Manises, Manises, Valencia
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital Lozano Blesa, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No